CLINICAL TRIAL: NCT06765577
Title: Prognostic Value of Finger Blood Pressure in Arteriovenous Fistula Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019/2459
Record Dates: First submitted 2024-11-12; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: End Stage Renal Disease; End-Stage Kidney Disease; Dialysis Access Dysfunction
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with End Stage Renal Failure undergoing Arteriovenous Fistula Creation (Experimental)
  Interventions: Other: Finger Blood Pressure Measurement

INTERVENTIONS:
Other: Finger Blood Pressure Measurement — Finger Blood Pressure Measurement were taken from three digits: the thumb (F1), the middle finger (F2), and the little finger (F3) from both arms.

SUMMARY:
The goal of this trial is to investigate the prognostic value of monitoring finger blood pressures (FBPs) in predicting the success of surgically created arteriovenous fistula (AVF) for patients with end stage renal disease. The main questions it aims to answer is:

- Can FBPs predict AVF maturation?

Participants will undergo FBP measurements at pre-op, immediately post-op, 4 weeks and 6 weeks post-AVF creation.

ELIGIBILITY:
Inclusion Criteria:

* Participants has documented Chronic Kidney Disease (CKD), determined by Glomerular Filtration Rate (GFR)
* Participant is recommended for renal replacement therapy based on clinical assessment of renal function as well as CKD staging, as documented in clinical notes.
* Haemodialysis was chosen as the most appropriate renal replacement therapy
* Participant is able to consent to the creation of an AVF in preparation for hemodialysis.
* Participant is able to adhere to follow-up assessments of AVF maturation, if applicable.

Exclusion Criteria:

* Subject had a previous AVF and is now undergoing surgery for another AVF creation
* Subject has amputation distal to AVF
* Subject is pregnant or planning to conceive
* Participants is unable to consent

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Correlation between AVF maturation and changes in Finger Blood Pressure measurements at baseline and immediately post-op | Within 24 hours
  To determine whether if there are any pattern in changes observed in FBP pre and post-creation that can be used for correlation to AVF maturation.

SECONDARY OUTCOMES:
Correlation between AVF maturation and changes in Finger Blood Pressure measurements across other timepoints | Until 6 weeks post-operation
  To determine whether changes in FBP across time points (pre-op, post-op, 4 weeks and 6 weeks post-op) is correlated with AVF maturation

CONTACTS AND LOCATIONS:
Overall Officials: Tze Tec Chong, MBBS, RPVI, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, SG, Singapore

IPD SHARING:
Plan to Share IPD: No
Personal Data Protection Act

REFERENCES:
- [Background] McGrogan DG, Maxwell AP, Khawaja AZ, Inston NG. Current tools for prediction of arteriovenous fistula outcomes. Clin Kidney J. 2015 Jun;8(3):282-9. doi: 10.1093/ckj/sfv019. Epub 2015 Apr 2. PMID 26034589
- [Background] Lee KG, Chong TT, Goh N, Achudan S, Tan YL, Tan RY, Choong HL, Tan CS. Outcomes of arteriovenous fistula creation, effect of preoperative vein mapping and predictors of fistula success in incident haemodialysis patients: A single-centre experience. Nephrology (Carlton). 2017 May;22(5):382-387. doi: 10.1111/nep.12788. PMID 27042772
- [Background] Alfano G, Fontana F, Cappelli G. Noninvasive Blood Pressure Measurement in Maintenance Hemodialysis Patients: Comparison of Agreement between Oscillometric and Finger-Cuff Methods. Nephron. 2017;136(4):309-317. doi: 10.1159/000457812. Epub 2017 May 4. PMID 28468005